CLINICAL TRIAL: NCT06195293
Title: Anti-cancer Neoantigen Polypeptide Vaccine to Treat Advanced Solid Tumors: Phase I Clinical Trial
Brief Title: Anti-cancer Neoantigen Polypeptide Vaccine to Treat Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZVACCINE-POLYPEPTIDE-021
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Solid Tumor, Adult
Keywords: Solid Tumor; Polypeptide Vaccine; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-cancer Neoantigen Polypeptide Vaccine (Experimental): Anti-cancer neoantigen polypeptide vaccine will be produced to treat advanced solid tumors.
  Interventions: Biological: Neoantigen Polypeptide Vaccine

INTERVENTIONS:
Biological: Neoantigen Polypeptide Vaccine — Deliver neoantigen polypeptide vaccine into patients for anti-ancer therapy.

SUMMARY:
The WES and RAN-seq will be performed to identify and verify neoantigens and appropriate polypeptide sequences will be verified, manufactured and protected for vaccine production by multiple in vitro and in vivo studies. Clinical studies will be performed to test anti-cancer function of the polypeptide vaccine for immunotherapy of human cancer patients. In this phase I study, the safety, tolerance, and preliminary efficacy of the polypeptide vaccine immunotherapy on human cancers will firstly be evaluated.

DETAILED DESCRIPTION:
1. Choose appropriate patients with advanced solid cancers, with written consent for this study;
2. Perform biopsy to get fresh sample for DNA/RNA-seqencings and bioinformatics analysis;
3. Produce appropriate polypeptide vaccine for human use and deliver the vaccine into selected patients via local injections, and follow up closely to collect related results as required;
4. To enhance the killing capability, cotreatment the patients with PD1/PDL1/CTLA4 antibodies may be applied;
5. Evaluate the clinical results as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced cancer; 2. Life expectancy >12 weeks; 3. Adequate heart, lung, liver, kidney, and blood function; 4. Available high quality vaccine for human use; 5. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

-

Exclusion Criteria:

1. Had accepted gene therapy before;
2. Severe virus infection such as HBV, HCV, HIV, et al;
3. Known HIV positivity;
4. Active infectious disease related to bacteria, virus,fungi,et al;
5. Other severe diseases that the investigators consider not appropriate;
6. Pregnant or lactating women;
7. Systemic steroid treatment (greater than or equal to 0.5 mg prednisone equivalent/kg/day);
8. Other conditions that the investigators consider not appropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2037-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicity | Six months
  A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the vaccine, which is irreversible, or life threatening or hematologic or non-hematologic Grade 3-5.

SECONDARY OUTCOMES:
Percent of Patients with best response as either complete remission or partial remission. | Six months
  Response rates will be estimated as the percent of patients whose best response is either complete remission or partial remission by combining the data from the patients. To compare with historical data, a 95% confidence interval will be calculated for the response rate.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD, PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, China